CLINICAL TRIAL: NCT03563378
Title: Effects of Intraoperative Normal Saline vs Lactated Ringer on Outcomes in Pediatric Liver Transplantation: A Double-blind Randomized Trial
Brief Title: Effects of Intraoperative Normal Saline vs Lactated Ringer on Outcomes in Pediatric Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-162
Record Dates: First submitted 2018-05-21; First posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Biliary Atresia Intrahepatic Syndromic Form
MeSH Terms: interventions — Ringer's Lactate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactated ringers solution (Experimental): Participants in this group will receive Lactated Ringer's solution during the intraoperative period.
  Interventions: Drug: Lactated Ringer
- Normal saline solution (Experimental): Participants in this group will receive Normal saline solution during the intraoperative period.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lactated Ringer — Patients will be administered Lactated Ringer's solution for intraoperative fluid management.
  Arms: Lactated ringers solution
Drug: Normal saline — Patients will be administered normal saline for intraoperative fluid management.
  Arms: Normal saline solution

SUMMARY:
Lactated Ringer(LR) has been extensively used to maintain and replace intravascular volume in a variety of anesthetic procedures. However, the utility of LR in pediatric with hepatic failure undergoing liver transplantation is unclear, because addition of exogenous lactate may increase lactate concentration. In addition,large amounts of normal saline(NS) which does not contain lactate can induce a hyperchloremic metabolic acidosis and have been asociated with adverse effects on kidney injury, coagulation, and death. Accordingly, the investigators performed a double-blinded randomized trial comparing the effects of intraoperative NS or LR on outcomes in pediatric receiving Liver transplantation.

ELIGIBILITY:
Criteria

Inclusion Criteria:

1. Pediatric patients between the age of 3 month and 6 years
2. Scheduled for living donor liver transplantation

Exclusion Criteria:

1. Re-transplantation
2. Combined liver and kidney transplantation
3. Congenital heart disease
4. Refused to participate the study

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2018-07-28 (Estimated); Primary Completion 2020-05-27 (Estimated); Study Completion 2020-05-27 (Estimated)

PRIMARY OUTCOMES:
Change in lactate level of the lactated ringer group compared to the normal saline group | up to 3 days after surgery
  Baseline serum lactate will be measured after randomization and again after surgery, then every 24 hours for 72 hours

SECONDARY OUTCOMES:
Length of mechanical ventilation | up to 30 days after surgery
  Length of mechanical ventilation in ICU measured in hours
ICU stay | up to 30 days after surgery
  Days spend in ICU within 30 days
30 day mortality | up to 30 days after surgery
  Patient mortality during the first 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: qi lu, Dr., Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided